CLINICAL TRIAL: NCT00984035
Title: Investigation of Germline Genetic Determinants and Early Biomarkers of Cisplatin-Related Nephrotoxicity
Brief Title: Investigation of Cisplatin-Related Kidney Toxicity
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: American Society of Clinical Oncology (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-135-B
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Biomarkers; Blood Specimen Collection; DNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Blood Serum/Plasma Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospecitive Analysis: Patients currently receiving cisplatin as treatment for their cancer.
  Interventions: Other: urine samples (biomarkers); Other: blood samples (biomarkers); Other: blood sample (DNA)
- Restrospective Analysis: Patients that have previously received cisplatin as treatment for their cancer.
  Interventions: Other: blood sample (DNA)

INTERVENTIONS:
Other: urine samples (biomarkers) — Urine samples collected prior to first dose of cisplatin, after each dose of cisplatin, and within 35 days of the last dose.
  Groups: Prospecitive Analysis
Other: blood samples (biomarkers) — blood samples collected prior to first dose of cisplatin, after each dose of cisplatin, and within 35 days of the last dose.
  Groups: Prospecitive Analysis
Other: blood sample (DNA) — Blood sample collected for DNA analysis at anytime while on-study.

SUMMARY:
The purpose of this study is to identify novel biomarkers of kidney injury in patients receiving cisplatin.

This study will also collect DNA for future analysis.

DETAILED DESCRIPTION:
This study will look for novel biomarkers of kidney injury in patients receiving cisplatin in patients currently receiving cisplatin.

DNA will be collected both prospectively and retrospectively (from patients that have previously received cisplatin.

ELIGIBILITY:
Prospective Analysis Group

Inclusion Criteria:

* Patients about to receive intravenous cisplatin for the first time as part of cancer chemotherapy.
* Aged 18 years and older.
* Ability to understand and willingness to sign a written consent document.
* Patients may be receiving cisplatin in combination with other chemotherapeutic agents.
* Patients may be receiving cisplatin in the context of another clinical trial.

Exclusion Criteria:

* Prior receipt of cisplatin.
* Patients on dialysis or other renal replacement therapy prior to starting cisplatin.
* Uncontrolled hypo- or hyperthyroidism (patients on chronic stable doses of thyroid replacement medication are eligible).

Retrospective Analysis Group

Inclusion Criteria:

* Patients that have previously received intravenous cisplatin as part of cancer chemotherapy.
* Aged 18 years and older.
* Ability to understand and willingness to sign a written consent document.
* Patients that received cisplatin in combination with other chemotherapeutic agents are eligible.
* Patients that received cisplatin in the context of a clinical trial are eligible.

Exclusion Criteria:

* Unable or unwilling to submit to a one-time blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving anti-cancer treatment with cisplatin (or previously treated with cisplatin) at a participating academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in urine biomarker (NGAL) after cisplatin | while on drug and up to 35 days after end of treatment

SECONDARY OUTCOMES:
Change in blood and urine cystatin C | while on drug and up to 35 days after end of treatment
Change in blood NGAL while receiving cisplatin | while on drug and up to 35 days after end of treatment
Genetic markers of kidney toxicity | while on drug and up to 35 days after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter H O'Donnell, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States